CLINICAL TRIAL: NCT03648931
Title: Qualitative Assessment of Acceptability of Vaginal Ring (VR) and Oral Pre-exposure Prophylaxis (PrEP) Use During Pregnancy and Breastfeeding
Brief Title: Microbicide/PrEP Acceptability Among Mothers and Male Partners in Africa
Acronym: MAMMA
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-041; UM1AI068633 (NIH); UM1AI068615 (NIH); UM1AI106707 (NIH); 38161 (Other: DAIDS)
Record Dates: First submitted 2018-08-02; First posted 2018-08-28 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2021-06

CONDITIONS: HIV Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant or Breastfeeding Women: No actual intervention is planned. A single focus group discussion (FGD) with community members in the same group assignment will be conducted to assess study outcome measures.
  Interventions: Behavioral: Focus Group Discussion (FGD)
- Male Partners: No actual intervention is planned. A single focus group discussion (FGD) with community members in the same group assignment will be conducted to assess study outcome measures.
  Interventions: Behavioral: Focus Group Discussion (FGD)
- Grandmothers: No actual intervention is planned. A single focus group discussion (FGD) with community members in the same group assignment will be conducted to assess study outcome measures.
  Interventions: Behavioral: Focus Group Discussion (FGD)
- Key Informants: No actual intervention is planned. A single in-depth interview (IDI) will be conducted to assess study outcome measures.
  Interventions: Behavioral: In-depth Interview (IDI)

INTERVENTIONS:
Behavioral: Focus Group Discussion (FGD) — No actual intervention is planned. A single focus group discussion (FGD) with community members in the same group assignment will be conducted to assess study outcome measures. In particular, the FGDs will focus on:
  * Perceptions of taboos and acceptable and/or typical practices during pregnancy, childbirth and breastfeeding
  * Perceptions of HIV risk during pregnancy and breastfeeding
  * Perceived role of male partners during pregnancy and breastfeeding
  * Main challenge(s) perceived with VR and oral PrEP use during pregnancy and breastfeeding
  * Main factor(s) perceived to facilitate VR and oral PrEP use during pregnancy and breastfeeding
  * Willingness to join a VR and/or oral PrEP study during pregnancy and breastfeeding
  Groups: Grandmothers; Male Partners; Pregnant or Breastfeeding Women
Behavioral: In-depth Interview (IDI) — No actual intervention is planned. A single in-depth interview (IDI) will be conducted to assess study outcome measures, focusing on the following topics:
  * Perceptions of taboos and acceptable and/or typical practices during pregnancy, childbirth and breastfeeding
  * Perceptions of HIV risk during pregnancy and breastfeeding
  * Perceived role of male partners during pregnancy and breastfeeding
  * Main challenge(s) perceived with VR and oral PrEP use during pregnancy and breastfeeding
  * Main factor(s) perceived to facilitate VR and oral PrEP use during pregnancy and breastfeeding
  * How others in their professional and social networks and communities would view the VR and/or oral PrEP use by pregnant and breastfeeding women
  Groups: Key Informants

SUMMARY:
The MTN-041 study is a multi-site exploratory study using focus group discussions (FGDs) and in-depth interviews (IDIs) to identify individual, interpersonal, social and cultural factors that may affect potential uptake of two safe and effective HIV prevention products, the monthly dapivirine (DPV) vaginal ring (VR) and daily oral pre-exposure prophylaxis (PrEP), by pregnant and breastfeeding women in Africa.

DETAILED DESCRIPTION:
MTN-041 is an exploratory study primarily designed to identify individual, interpersonal, social and cultural factors that may affect potential uptake of two safe and effective HIV prevention products, the monthly DPV VR and daily oral PrEP, in a vulnerable yet seldom-studied population, pregnant and breastfeeding women. MTN-041 will utilize FGDs and IDIs to elicit community and health professional perceptions about vaginal practices, sexual activity, use of medicines, and HIV risk during pregnancy or breastfeeding, including how these perceptions may affect pregnant and breastfeeding women's acceptability of using intravaginal products and oral medications like the DPV VR and Truvada oral tablet.

The MTN-041 study population will consist of HIV-uninfected women 18-40 years old who are currently or were recently (within two years) pregnant or breastfeeding, men aged 18 years or older whose partners are currently or were recently (within two years) pregnant or breastfeeding, grandmothers whose daughters or daughters-in-law are currently or were recently (within two years) pregnant or breastfeeding, and key informants (KIs), which include: health care professionals (HCPs), traditional birth attendants (TBAs), providers of family planning, antenatal, and traditional health services to women, providers of other social services to women, and community leaders.

Up to 60 men and women will be selected at each site for participation in this study, for a maximum total of 240 study participants. This includes up to 50 FGD participants (currently or recently pregnant or breastfeeding women, male partners of women who are currently or were recently pregnant or breastfeeding, and grandmothers with currently or recently pregnant or breastfeeding daughters/daughters-in-law) and up to 10 KIs selected at each site, for a maximum total of 200 FGD participants and 40 KIs enrolled across all sites.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent in one of the study languages.
2. Able and willing to complete the required study procedures.

   For currently or recently pregnant or breastfeeding women:
3. Between the ages of 18 to 40 years old (inclusive) at Enrolment, verified per site standard operating procedures (SOPs).
4. Currently or recently (within two years) pregnant or breastfeeding (by self-report).

   For male partners:
5. Aged 18 years or older at Enrolment, verified per site SOPs.
6. Identifies as a primary sexual partner of a woman who is currently or was recently (within two years) pregnant or breastfeeding.

   For grandmothers:
7. Aged 18 years or older at Enrolment, verified per site SOPs.
8. Identifies as the maternal or paternal grandmother of a daughter or daughter-in-law who is currently or was recently (within two years) pregnant or breastfeeding.

   Note: The term "daughter-in-law" includes women who are/were not married to their male partner during or after pregnancy.

   For service provider KIs:
9. Aged 18 years or older at Enrolment, verified per site SOPs.
10. Currently working as a clinician (e.g., obstetrician, nurse, pharmacist, etc.), traditional care provider (e.g., TBA, healer, midwife, etc.), social service provider (e.g., social worker, family planning counselor, etc.) or community health worker in one of the study countries, verified per site SOPs.
11. Experienced in providing services to pregnant and/or breastfeeding women.

    For community leader KIs:
12. Aged 18 years or older at Enrolment, verified per site SOPs.
13. Currently acting in a community leadership role (e.g., local chief, religious leader, etc.).

Exclusion Criteria:

1. Has any condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
2. For currently or recently pregnant or breastfeeding women: known HIV-positive status, verified per recent health record (e.g., health passport, ante-natal book, HIV test card, or similar document) or by self-report if health record(s) not available.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The MTN-041 study population will consist of HIV-uninfected women 18-40 years old who are currently or were recently (within two years) pregnant or breastfeeding, men aged 18 years or older whose partners are currently or were recently (within two years) pregnant or breastfeeding, grandmothers whose daughters or daughters-in-law are currently or were recently (within two years) pregnant or breastfeeding, and key informants (KIs), which include: health care providers (HCPs), traditional birth attendants (TBAs), providers of family planning, antenatal, and traditional health services to women, providers of other social services to women, and community leaders.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Acceptability of VR during pregnancy and breastfeeding, including willingness to use the VR or support its use | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews
Acceptability of oral PrEP during pregnancy and breastfeeding, including willingness to use oral PrEP or support its use | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews

SECONDARY OUTCOMES:
Product preferences during pregnancy and breastfeeding | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews
Sexual activity and contraceptive use during pregnancy and breastfeeding | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews
Perceptions of HIV risk during pregnancy and breastfeeding | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews
Community beliefs and practices related to pregnancy and breastfeeding, including use of oral medications and intravaginal products | 3-6 months during Q2/Q3 2018
  Focus group discussions and key informant in-depth interviews

CONTACTS AND LOCATIONS:
Overall Officials: Ariane van der Straten, PhD, MPH, Study Chair — Women's Global Health Imperative Program, RTI International
Locations (4):
- Blantyre Clinical Research Site, Blantyre, Malawi
- Wits Reproductive Health and HIV Institute (WRHI) Clinical Research Site, Johannesburg, South Africa
- Makerere University - Johns Hopkins University (MU-JHU) Research Collaboration Clinical Research Site, Kampala, Uganda
- Zengeza Clinical Research Site, Harare, Zimbabwe

REFERENCES:
- [Result] van der Straten A, Ryan JH, Reddy K, Etima J, Taulo F, Mutero P, Taylor J, Piper J, Musara P; MTN-041/MAMMA Study Team. Influences on willingness to use vaginal or oral HIV PrEP during pregnancy and breastfeeding in Africa: the multisite MAMMA study. J Int AIDS Soc. 2020 Jun;23(6):e25536. doi: 10.1002/jia2.25536. PMID 32524700
- [Result] Flax VL, Hawley I, Ryan J, Chitukuta M, Mathebula F, Nakalega R, Seyama L, Taulo F, van der Straten A; MTN-041/MAMMA Study Team. After their wives have delivered, a lot of men like going out: Perceptions of HIV transmission risk and support for HIV prevention methods during breastfeeding in sub-Saharan Africa. Matern Child Nutr. 2021 Apr;17(2):e13120. doi: 10.1111/mcn.13120. Epub 2020 Dec 15. PMID 33325126